CLINICAL TRIAL: NCT04487665
Title: Oral Manifestations of COVID-19: a Multicentre Observational Study
Brief Title: Oral Manifestations of Coronavirus Disease 2019(COVID-19) :a Multicentre Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dina mounir elkady, lecturer at conservative department, Cairo University
Other Study IDs: 8791
Record Dates: First submitted 2020-07-21; First posted 2020-07-27 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- positive COVID-19: patient diagnosed by nasopharyngeal positive COVID-19

SUMMARY:
online questionnaire will be distributed in different country to detect the oral change in patient diagnosed with COVID-19

DETAILED DESCRIPTION:
an online survey will be performed through google form. Investigators in different country will share the questionnaire with patient diagnosed positive COVID-19.

data collected will be statically analyse to detect the oral picture of the virus.

ELIGIBILITY:
Inclusion Criteria:

* positive COVID-19

Exclusion Criteria:

* children
* patient not confirmed by swab

Ages: 18 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: patient with no previous serious illness - from different country
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-09-15 (Estimated); Primary Completion 2020-11-15 (Estimated); Study Completion 2020-12-15 (Estimated)

PRIMARY OUTCOMES:
oral ulcer | through study completion, an average of 1 month
  number of patient with oral ulcer

SECONDARY OUTCOMES:
hyposalivation | through study completion, an average of 1 month
  change in salivary flow

IPD SHARING:
Plan to Share IPD: No
data will be on a private mail , no access will be provided except for principal investigator